CLINICAL TRIAL: NCT07104409
Title: Virtual Reality Hypnosis as Sedation During Oocyte Retrieval: Effect on Propofol Consumption: a Randomized Study (VRH-IVF)
Brief Title: Virtual Reality Hypnosis as Sedation During Oocyte Retrieval: Effect on Propofol Consumption
Acronym: VRH-IVF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/24JUI/253; VRH-IVF (Registry Identifier: 2025/24JUI/253)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Oocyte Retrieval for IVF
Keywords: virtual reality; hypnosis; oocyte retrieval

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): sedation with remifentanil and propofol
- RVH group (Experimental): RVH session + sedation with remifentanil and propofol
  Interventions: Other: virtual reality hypnosis device

INTERVENTIONS:
Other: virtual reality hypnosis device — VRH group, in which patients will receive conventional sedation (remifentanil 0.1 mcg/kg/min and propofol 0.5 mg/kg if necessary) and a Virtual Reality headset with an environment chosen by the patient and hypnosis support with suggestions to reduce their anxiety.
  Arms: RVH group

SUMMARY:
An egg retrieval is performed during an IVF course. This painful procedure is performed using sedation to ensure patient comfort. A combination of sedative and analgesic medications combined with local anesthesia (paracervical block) is used. Propofol, the intravenous anesthetic of choice (rapid-acting and short-acting), and remifentanil (an ultra-short-acting opioid analgesic) are generally combined. The potential impact of these agents used for egg retrieval on egg fertilization and embryo quality is of interest. Indeed, certain drugs such as propofol could accumulate in the follicular fluid. The few studies conducted to date show contradictory results. While a harmful effect appears to be reported in experimental studies on mice, this effect is uncertain in clinical studies. Given this uncertainty, any method aimed at reducing propofol consumption in this context may be of interest. Virtual reality hypnosis (VRH) is a digital tool that has already been shown to be effective in reducing preoperative anxiety during oocyte retrieval. Furthermore, VRH has also demonstrated analgesic effects.

The primary objective of this study is to compare VRH with a control group (usual sedation) on propofol consumption during oocyte retrieval.

Secondary objectives are to compare preoperative anxiety, APAIS score, catastrophizing score, remifentanil consumption, intra- and/or post-operative nausea and vomiting, post-procedural analgesic consumption, time perception during the procedure, fertilization parameters, and pregnancy rate at 12 weeks. The degrees of absorption, dissociation, immersion, and presence for the VRH group will also be noted.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, controlled interventional study that will include 72 patients. Patients will be randomized into two groups: a Control group, in which patients will receive conventional sedation (remifentanil 0.1 mcg/kg/min and propofol 0.5 mg/kg if necessary) during the retrieval, and an RVH group, in which patients will receive conventional sedation (remifentanil 0.1 mcg/kg/min and propofol 0.5 mg/kg if necessary) and a Virtual Reality headset with an environment chosen by the patient and hypnosis support with suggestions to reduce their anxiety. To be included, patients must have undergone egg retrieval as part of their IVF at the Cliniques universitaires Saint-Luc, be French-speaking, have undergone simple IVF or ICSI IVF, and must not be undergoing long-term psychotherapeutic treatment or taking psychotropic medications. They must also have given their free, informed and written consent signed by the investigator and the patient in the days preceding the intervention. Patients with morbid obesity, blindness and/or deafness and with a history contraindicating the use of anti-inflammatory drugs will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* egg retrieval as part of their IVF at the Cliniques universitaires Saint-Luc,
* to be French-speaking,
* simple IVF or ICSI IVF
* 18-42 yrs

Exclusion Criteria:

* morbid obesity
* blindness and/or deafness
* history contraindicating the use of anti-inflammatory drugs
* long-term psychotherapeutic treatment or taking psychotropic medications.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only people who has oocyte retrieval for IVF
Enrollment: 72 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study is to compare VRH with a control group (usual sedation) on propofol consumption during the procedure. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Roelants, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the study will not be made available due to lack of consent for data sharing.

REFERENCES:
- [Background] Rousseaux F, Panda R, Toussaint C, Bicego A, Niimi M, Faymonville ME, Nyssen AS, Laureys S, Gosseries O, Vanhaudenhuyse A. Virtual reality hypnosis in the management of pain: Self-reported and neurophysiological measures in healthy subjects. Eur J Pain. 2023 Jan;27(1):148-162. doi: 10.1002/ejp.2045. Epub 2022 Oct 24. PMID 36196745
- [Background] Pirard C, Laurent P, Wyns C, Giudice MG, Watremez C, Momeni M, Roelants F. Impact of virtual reality with or without hypnosis before oocyte retrieval: A randomised study. Complement Ther Med. 2025 Mar;88:103125. doi: 10.1016/j.ctim.2024.103125. Epub 2025 Jan 3. PMID 39756588
- [Background] Matsota P, Sidiropoulou T, Vrantza T, Boutsikou M, Midvighi E, Siristatidis C. Comparison of Two Different Sedation Protocols during Transvaginal Oocyte Retrieval: Effects on Propofol Consumption and IVF Outcome: A Prospective Cohort Study. J Clin Med. 2021 Mar 1;10(5):963. doi: 10.3390/jcm10050963. PMID 33804575